CLINICAL TRIAL: NCT02856061
Title: Tracking Intervention Effects With Eye Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Simons Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1106008625a; 383661 (Other Grant/Funding Number: Simons Foundation Autism Research Initiative)
Record Dates: First submitted 2016-07-12; First posted 2016-08-04 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

ARMS (3):
- PRT (Other): Children with ASD who are currently receiving PRT treatment.
  Interventions: Behavioral: Pivotal Response Treatment
- Wait List / Non-Treatment Control (No Intervention): Children with ASD who are not currently receiving PRT treatment.
- Typically Developing (No Intervention): Children without ASD or developmental delay.

INTERVENTIONS:
Behavioral: Pivotal Response Treatment — Pivotal response treatment (PRT) is an empirically validated behavioral treatment for individuals with ASD that has its foundation in principles of Applied Behavioral Analysis. It was designed to improve social communication skills by addressing core deficits in social motivation or pivotal responses. By working specifically with each child's natural motivations, PRT focuses on naturalistic, functional skills, as opposed to rote skills. In this study, participants randomized to the PRT group will receive 6 hours of direct PRT, across three sessions per week, provided by Dr. Ventola's clinical team. Parents will have an additional one-hour session per week focused on PRT parent training using a practice-with-feedback model. Specific intervention goals in our target population include: Speech to respond to inquiries, Speech to inquire, Speech to comment, Reciprocal conversation, Monitor nonverbal information, and Perspective taking.
  Arms: PRT

SUMMARY:
This pilot study examines concurrent and predictive relationships between eye tracking and clinical outcomes during a 16-week behavioral intervention (PRT) for children with ASD. Eye tracking will be comprised of both laboratory-based measures (using a commercial eye-tracking system) as well as home-based measures (using tablet-based eye tracking systems). The major goals of this study are both to improve our understanding of the potential role of eye tracking in clinical trials and to advance technologies that may further improve the sensitivity, robustness, accessibility, and ultimate utility of eye tracking methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 4-7 years diagnosed previously with ASD and meet criteria for ASD when characterized by our research team, English is a language spoken in the family, and Full-scale IQ>50. Participants must also complete laboratory and home-based eye tracking sessions, with success determined by the Principal Investigator.

Exclusion Criteria:

* Individuals will be excluded from participation based on the presence of

  1. a physical or neurological disorder (e.g., cerebral palsy) which is likely to impact development and learning, as intervention procedures for these individuals may need to be modified beyond the standard approach to address more complex developmental needs,
  2. hearing loss or other severe sensory impairment,
  3. history of significant head trauma or serious brain or psychiatric illness,
  4. parents/caregivers who do not speak fluent English,
  5. parents/caregivers who have previous training in PRT
  6. individuals who must be excluded from eye tracking. These families will be offered the treatment clinically (i.e., fee-based), and they will be given referrals to outside agencies offering the treatment as well.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Laboratory Eye Tracking Measuring Longitudinal Change | 16 Weeks
  A comprehensive laboratory eye-tracking battery will be administered to participants before, at midpoint, and at the end of a 16-week period to assess change over the course of treatment.
Home-Based Eye Tracking | 16 Weeks
  Participants will also receive a tablet equipped with eye-tracking paradigms specifically designed for continuous monitoring in homes. Caregivers will be asked to complete a brief questionnaire
Longitudinal Change in Autism Symptom Severity | 16 Weeks
  Clinical assessments and caregiver surveys will be administered at baseline. A subset of measures will be administered again post-study. Assessments include the Autism Diagnostic Observation Schedule™ Second Edition (ADOS™-2), Autism Diagnostic Interview™ Revised (ADI™-R), Social Responsiveness Scale™ (SRS™), Repetitive Behaviors Scale - Revised (RBS-R), Differential Ability Scales®-II (DAS-II®), Vineland Adaptive Behavior Scales™ Second Edition (Vineland™-II), and the Child Behavior Checklist (CBCL).

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Shic, PhD, Principal Investigator — Yale University; Pamela Ventola, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States